CLINICAL TRIAL: NCT03562728
Title: Assessing the Functional Impact of Progressive Rehabilitation Therapy in Patients With Advanced Lung Disease Requiring Lung Transplantation or ECMO- Bridge to Transplant
Brief Title: Progressive Rehabilitation Therapy in Patients With Advanced Lung Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Irina Timofte, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00080970
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Advanced Lung Disease; Lung Transplant; Extracorporeal Membrane Oxygenation
Keywords: Transplant; ECMO; Sarcopenia; Deconditioning; Physical therapy
MeSH Terms: conditions — Sarcopenia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ECMO- Bridge to Transplant (Active Comparator): Interventions: MRP+MNES(neuromuscular electric stimulation).Patients in the treatment arm will receive additional physical therapy(arm and leg exercises, using light weight machines, hand weights, or rubber bands, exercise machines such as portable arm or seated bikes) as well as therapy with an electric stimulator device. This device uses weak electric impulses to involuntarily exercise the muscles(one-two sessions a day).Four muscle groups(quadriceps and dorsiflexors bilaterally) will be stimulated using surface electrodes .In addition, patients in the experimental group will receive nutrition supplementation with essential amino acids 3 times a day in their feeding to prevent muscle breakdown and promote positive nitrogen balance.
  Interventions: Device: MRP and NMES(neuromuscular electric stimulation)
- ECMO- Bridge to Transplant Control Group (Other): Interventions: standard of care
  Patients are not going to receive any additional intervention.
  Interventions: Other: Standard of Care
- Transplant (Active Comparator): Interventions: MRP+MNES(neuromuscular electric stimulation).Patients in the treatment arm will receive additional physical therapy(arm and leg exercises, using light weight machines, hand weights, or rubber bands, exercise machines such as portable arm or seated bikes) as well as therapy with an electric stimulator device. This device uses weak electric impulses to involuntarily exercise the muscles(one-two sessions a day).Four muscle groups(quadriceps and dorsiflexors bilaterally) will be stimulated using surface electrodes .In addition, patients in the experimental group will receive nutrition supplementation with essential amino acids 3 times a day in their feeding to prevent muscle breakdown and promote positive nitrogen balance.
  Interventions: Device: MRP and NMES(neuromuscular electric stimulation)
- Transplant Control Group (Other): Interventions: standard of care.
  Patients are not going to receive any additional intervention.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: MRP and NMES(neuromuscular electric stimulation) — nutrition supplementation includes addition of essential amino acids 3 times a day to feeding
  Other Names: Dietary Supplement(NS)
  Arms: ECMO- Bridge to Transplant; Transplant
Other: Standard of Care — Patients in the control group are going to receive standard of care
  Arms: ECMO- Bridge to Transplant Control Group; Transplant Control Group

SUMMARY:
The International Society of Heart and Lung Transplantation Registry data shows that there is a growing population of critically ill patients with advanced lung disease undergoing lung transplantation.

The goal of our study is to evaluate the role of intensive physical therapy for patients with advanced lung disease requiring transplant or ECMO(extracorporeal membrane oxygenation)- bridge to transplant with emphasis on the restoration of functional independence and prevention of functional declines after lung transplantation.

The project is a designed as a randomized prospective research study investigating the impact of a multi-modal rehabilitation program(MRP), which incorporates neuromuscular electric stimulation(NMES), strength and mobility training, and nutritional supplementation(NS) in ameliorating the loss of muscle mass and strength, and lower extremity balance, strength and coordination that will decrease time on the ventilator or ECMO, stay in the ICU and hospital.

DETAILED DESCRIPTION:
Intensive rehabilitation is recognized as an essential component to successful outcomes for post procedure recovery after a major cardio-thoracic procedure. The investigators propose a unique multi-modal rehabilitation program (MRP) that combines a step-up physical therapy protocol with neuromuscular electric stimulation (NMES), nutritional supplementation (NS), occupational therapy and pulmonary rehabilitation techniques to achieve improved functional outcomes for advanced lung disease patients requiring transplantation or ECMO-bridge to transplant. The investigators hypothesized that a progressive rehabilitation program, incorporating neuromuscular electric stimulation, strength and balance training, and nutritional supplementation with essential amino acids will reduce sarcopenia and loss of functional mobility in patients with advanced lung disease requiring transplantation or ECMO-bridge to transplant.

The purpose of this study is to determine the effectiveness of a progressive rehabilitation program, which incorporates neuromuscular electric stimulation, strength and mobility training, and nutritional supplementation in ameliorating 1) the loss of muscle mass and strength, and lower extremity balance, strength and coordination, 2) time on the ventilator or ECMO, stay in the intense care unit and hospital, and 3) return home and quality of life compared to usual ICU care.

The investigators propose a prospective, randomized interventional trial assessing the effectiveness of the program in decreasing adverse post-transplant outcomes compared to usual care. All advanced lung disease patients listed for transplantation or requiring ECMO cannulation will be screened for this study according to the inclusion and exclusion criterion. The patients will be randomized to either the treatment arm or usual care within 72 hours after the procedure (transplant or ECMO cannulation if patient requires ECMO-bridge to transplant). All groups of patients will undergo an initial global assessment of functional capabilities after listing for lung transplantation and then again within 72 hours after cardio-thoracic procedure (transplant or ECMO cannulation). Patients in the treatment arm will receive additional physical therapy that include: arm and leg exercises, using light weight machines, hand weights, or rubber bands, exercise machines such as portable arm or seated bikes. The treatment group will receive exercise therapy plus therapy with an electric stimulator device. This device uses weak electric impulses to involuntarily exercise the muscles (one-two sessions a day, with each session starting off at 10 minutes, then increasing to a maximum of 30 minutes). Subjects receiving the intervention will receive daily treatment using the neuromuscular electric stimulation unit. Four muscle groups (quadriceps and dorsiflexors bilaterally) will be stimulated using 3x5 inch surface electrodes (quadriceps) and 2x4 inch (dorsiflexors). In addition, patients in the experimental group will receive nutrition supplementation with essential amino acids 3 times a day in their feeding to prevent muscle breakdown and promote positive nitrogen balance. Comprehensive re-assessments are repeated on a weekly basis and the therapy will be adjusted to the patient's clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Advanced lung disease requiring lung transplantation
* Advanced lung disease requiring ECMO bridge to lung transplantation
* Patient or legally authorized representative are able to provide written or witnessed verbal consent.

Exclusion Criteria:

* Unable to obtain consent from patient or family member
* Advanced lung disease but not transplant candidate due to other comorbidities
* Patient is deemed unsafe for rehabilitation by the transplant physician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Global muscle strength | 14 days
  Muscle group strength is obtained using hand held dynamometer
Mobility status | 14 days
  Mobility status is assessed with 6 minute walk distance
Muscle mass | 14 days,
  Muscle mass measurement of lower extremity muscle volume using ultrasound scan or computer tomography

SECONDARY OUTCOMES:
Time on the ventilator or ECMO | 14 days, 1 month
  Measured as ECMO or ventilator days
Stay in the ICU and hospital | 14 days, 1,3month
  Measured as days in the ICU and hospital

CONTACTS AND LOCATIONS:
Overall Officials: Irina Timofte, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Information will be shared only with the investigators that are actively involved in the study

REFERENCES:
- [Background] Downs AM. Physical therapy in lung transplantation. Phys Ther. 1996 Jun;76(6):626-42. doi: 10.1093/ptj/76.6.626. PMID 8650277
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Vogiatzis I, Terzis G, Nanas S, Stratakos G, Simoes DC, Georgiadou O, Zakynthinos S, Roussos C. Skeletal muscle adaptations to interval training in patients with advanced COPD. Chest. 2005 Dec;128(6):3838-45. doi: 10.1378/chest.128.6.3838. PMID 16354852
- [Background] Williams TJ, Patterson GA, McClean PA, Zamel N, Maurer JR. Maximal exercise testing in single and double lung transplant recipients. Am Rev Respir Dis. 1992 Jan;145(1):101-5. doi: 10.1164/ajrccm/145.1.101. PMID 1731570
- [Background] Vogiatzis I, Nanas S, Roussos C. Interval training as an alternative modality to continuous exercise in patients with COPD. Eur Respir J. 2002 Jul;20(1):12-9. doi: 10.1183/09031936.02.01152001. PMID 12166558
- [Background] Chambers DC, Yusen RD, Cherikh WS, Goldfarb SB, Kucheryavaya AY, Khusch K, Levvey BJ, Lund LH, Meiser B, Rossano JW, Stehlik J; International Society for Heart and Lung Transplantation. The Registry of the International Society for Heart and Lung Transplantation: Thirty-fourth Adult Lung And Heart-Lung Transplantation Report-2017; Focus Theme: Allograft ischemic time. J Heart Lung Transplant. 2017 Oct;36(10):1047-1059. doi: 10.1016/j.healun.2017.07.016. Epub 2017 Jul 19. No abstract available. PMID 28784324
- [Background] Alon G, V Smith G. Tolerance and conditioning to neuro-muscular electrical stimulation within and between sessions and gender. J Sports Sci Med. 2005 Dec 1;4(4):395-405. eCollection 2005 Dec. PMID 24501553